CLINICAL TRIAL: NCT00515450
Title: A Randomized, Controlled Clinical Study of GB-0998 for Treatment of Generalized Myasthenia Gravis
Brief Title: Efficacy and Safety Study of GB-0998 for Treatment of Generalized Myasthenia Gravis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Benesis Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0998-B1
Record Dates: First submitted 2007-08-10; First posted 2007-08-13 (Estimated); Last update posted 2010-07-30 (Estimated); Status verified 2010-07

CONDITIONS: Generalized Myasthenia Gravis
Keywords: Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis | interventions — Immunoglobulins, Intravenous; Plasmapheresis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Biological: GB-0998 (Intravenous immunoglobulin)
- 2 (Active Comparator)
  Interventions: Procedure: Plasmapheresis

INTERVENTIONS:
Biological: GB-0998 (Intravenous immunoglobulin)
  Other Names: Venoglobulin-IH
  Arms: 1
Procedure: Plasmapheresis
  Arms: 2

SUMMARY:
This randomized controlled, multi-center study will carry out to assess the efficacy of GB-0998 compared to plasmapheresis in the treatment of the generalized Myasthenia Gravis based on the changes in Quantitative Myasthenia Gravis score (QMG score) as primary endpoint, and in addition, to assess the safety of GB-0998

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as generalized myasthenia gravis
* Patients who are not controlled by current therapy and need plasmapheresis therapy
* Patients who have the high-dose steroid therapy for over a month in past years, and also who take steroid or immunosuppressant on the day of consent
* Patients who had not any dose increase or new dosing of steroid or immunosuppressant within 4 weeks prior to enrollment

Exclusion Criteria:

* Patients who received steroid pulse therapy, globulin therapy or plasmapheresis therapy within 12 weeks prior to enrollment
* Patients who had undergone thymectomy within 24 weeks prior to enrollment
* Patients with 3 points item in bulbar symptom of MG-ADL scale
* Patients with severe hepatic disorder, severe renal disorder or severe heat disorder
* Patients who have received treatment of malignant tumors
* Patients who have the anamnesis of shock or hypersensitivity to this drug
* Patients who have been diagnosed as hereditary fructose intolerance
* Patients who have the anamnesis of cerebral infarction or symptom of these diseases
* Patients who have been diagnosed as IgA deficiency in their past history
* Pregnant, lactating, and probably pregnant patients, and patients who want to become pregnant
* Patients who were administered other investigational drug within 12 weeks before consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2007-07; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Changes in QMG score | at 4 weeks

SECONDARY OUTCOMES:
Changes of QMG score, MG-ADL scale, anti-acetylcholine receptor antibody levels | from beginning of the treatment through 4th week

CONTACTS AND LOCATIONS:
Overall Officials: Masaharu Takamori, Director, Study Chair — Neurological Center Kanazawa-Nishi Hospital
Locations (1):
- Nagasaki University, Nagasaki, Nagasaki, Japan